CLINICAL TRIAL: NCT03778463
Title: Synovectomy Versus no Synovectomy in Primary Total Knee Arthrplasty : A Randomized Control Trial
Brief Title: Synovectomy in Primary Total Knee Arthrplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Saeed Younis, Principle investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12370677
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Arthroplasty, Replacement, Knee; Synovectomy
MeSH Terms: interventions — Synovectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Synovectomy (Experimental)
  Interventions: Other: Synovectomy
- No synovectomy (No Intervention)

INTERVENTIONS:
Other: Synovectomy — Removal of the synovium during total knee arthroplasty
  Arms: Synovectomy

SUMMARY:
The aim of total knee arthroplasty is to achieve best patient functional outcomes, improve patient pain score and satisfaction. Synovial proliferation is a common finding in arthritic knees. Surgeons can't decide if synovectomy is a crucial step in the operation. Studies didn't prove the clear benefits of synovectomy. We are aiming to perform a randomized clinical trial trying to reach the best evidence in that matter.

ELIGIBILITY:
Inclusion Criteria:

* patients with primary osteoarthritis undergoing primary total knee arthroplasty

Exclusion Criteria:

* Inflammatory arthritis
* Revision knee arthroplasty

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Functional outcome scores. e.g. knee society score (KSS) | one year
knee pain e.g. visual analogue score (VAS) score | immediate postoperative
Health related quality of life e.g. short form (SF12) scale | one year
Revision rate | one year
Reoperation rate | one year
Range of motion | immediate postoperative
Range of motion | 6 month
Range of motion | One year

SECONDARY OUTCOMES:
Postoperative blood loss | immediate postoperative
Postoperative hemoglobin level | immediate postoperative
  gram/dl
Infection rate | in first three month
Wound complications | in first 3 months
Number of patients requiring transfusion | immediate postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Saeed Younis, Dr., Principal Investigator — Ain Shams University; Amr Amal Elsayed Amin, Dr., Study Director — Ain Shams University; Wael Samir Osman, Professor, Study Chair — Ain Shams University
Locations (1):
- Ain Shams Univrsity, Cairo, Egypt